CLINICAL TRIAL: NCT00597584
Title: AFX01-14: A Phase 3, Randomized, Active-controlled, Open-label, Multi-center Study of the Safety and Efficacy of Peginesatide for the Maintenance Treatment of Anemia in Hemodialysis Patients Previously Treated With Epoetin
Brief Title: Safety & Efficacy of Peginesatide for Maintenance Treatment of Anemia in Participants With Chronic Kidney Disease on Hemodialysis
Acronym: EMERALD 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Affymax (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFX01-14; 2007-004153-28 (EudraCT Number)
Record Dates: First submitted 2008-01-10; First posted 2008-01-18 (Estimated); Results first posted 2012-07-30 (Estimated); Last update posted 2013-03-08 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Renal Failure; Chronic Kidney Disease; Anemia
Keywords: anemia; chronic kidney disease; CKD; chronic renal failure; CRF; dialysis; erythropoietin; EPO; erythropoiesis stimulating agent; ESA; Hematide™; hemodialysis; hemoglobin; Hb; Hgb; Omontys; peginesatide; red blood cell; red blood cell production
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic; Anemia | interventions — peginesatide; hematide; Epoetin Alfa; epoetin beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Peginesatide (Experimental)
  Interventions: Drug: peginesatide
- Epoetin (Active Comparator)
  Interventions: Drug: Epoetin alfa or Epoetin beta

INTERVENTIONS:
Drug: peginesatide — Participants received peginesatide by intravenous (IV) or subcutaneous (SC) injection once every 4 weeks. The starting dose was based on the participant's total weekly epoetin alfa or beta dose during the last week of the Screening Period; the first dose was administered one week after the last epoetin alfa or beta dose. Participants who received epoetin alfa or beta IV at the time of screening received peginesatide IV during the study, and participants who received epoetin alfa or beta SC at the time of screening received peginesatide SC during the study.
  The dose was adjusted to maintain hemoglobin levels in a target range of 10.0-12.0 g/dL and ± 1.5 g/dL from baseline during the Titration and Evaluation Periods, and 10.0-12.0 g/dL during the Long-Term Safety and Efficacy Period.
  Other Names: Omontys; Hematide; AF37702 Injection
  Arms: Peginesatide
Drug: Epoetin alfa or Epoetin beta — Participants continued to receive commercially available epoetin alfa or beta by intravenous or subcutaneous injection, at the same starting dose, frequency and route of administration as received during the last week of the Screening Period, with the first study dose of epoetin alfa or beta administered after randomization at Week 0.
  The dose was adjusted to maintain hemoglobin levels in a target range of 10.0-12.0 g/dL and ± 1.5 g/dL from baseline during the Titration and Evaluation Periods, and 10.0-12.0 g/dL during the Long-Term Safety and Efficacy Period.
  Other Names: Epogen; Neorecormon
  Arms: Epoetin

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of peginesatide in the maintenance treatment of anemia in participants on dialysis.

DETAILED DESCRIPTION:
Anemia associated with chronic kidney disease is due to several factors, primarily the inability of the diseased kidneys to produce adequate amounts of endogenous erythropoietin. Ancillary factors include the shortened lifespan of red blood cells, iron and other nutritional deficiencies, infection, and inflammation. The presence and severity of anemia are related to the duration and extent of kidney failure. Anemia is associated with increased mortality, increased likelihood of hospitalization, reduced cognitive function, and increased left ventricular hypertrophy and heart failure.

Erythropoiesis stimulating agents (ESAs) have been established as a treatment for anemia in chronic renal failure subjects, and have improved the management of anemia over alternatives such as transfusion. Peginesatide is a parenteral formulation developed for the treatment of anemia in patients with chronic kidney disease. Peginesatide binds to and activates the human erythropoietin receptor and stimulates erythropoiesis in human red cell precursors in a manner similar to other known erythropoiesis-stimulating agents.

Eligible participants were randomized in a 2:1 ratio to peginesatide administered once every 4 weeks or to continued treatment with epoetin administered 1-3 times each week, respectively. Total commitment time for this study was 4 weeks of screening followed by a minimum of 52 weeks of study treatment.

To evaluate the cardiovascular safety of peginesatide injection, a composite safety endpoint (CSE) was defined for use in prospectively planned analyses which combined cardiovascular safety data from the four Phase 3 peginesatide injection studies (NCT00598273, NCT00597753, NCT00598442, and NCT00597584). The CSE consisted of six events: death, stroke, myocardial infarction, and serious adverse events of congestive heart failure, unstable angina, and arrhythmia. An independent Event Review Committee (ERC) was used to provide blinded adjudication of potential CSE events.

ELIGIBILITY:
Inclusion Criteria

1. Participants with chronic renal failure on hemodialysis for ≥ 3 months prior to randomization.
2. On IV epoetin alfa or beta maintenance therapy continuously prescribed for a minimum of 8 weeks prior to randomization.
3. Four consecutive hemoglobin values with a mean ≥ 10.0 and ≤ 12.0 g/dL during the Screening Period.

Exclusion Criteria

1. Females who are pregnant or breast-feeding.
2. Known intolerance to any erythropoiesis stimulating agent or pegylated molecule or to all parenteral iron supplementation products.
3. Known bleeding or coagulation disorder.
4. Known hematologic disease or cause of anemia other than renal disease
5. Poorly controlled hypertension.
6. Evidence of active malignancy within one year prior to randomization.
7. Temporary (untunneled) dialysis access catheter.
8. A scheduled kidney transplant.
9. A scheduled surgery that may be expected to lead to significant blood loss.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 823 (Actual)
Dates: Start 2007-10; Primary Completion 2009-07 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President, Clinical Development, Study Director — Affymax
Locations (72):
- United States (36):
  - Research Facility, Phoenix, Arizona
  - Research Facility, Hot Springs, Arkansas
  - Research Facility, McGehee, Arkansas
  - Research Facility, Pine Bluff, Arkansas
  - Research Facility, Bakersfield, California
  - Research Facility, Glendale, California
  - Research Facility, Los Angeles, California
  - Research Facility, Riverside, California
  - Research Facility, Simi Valley, California
  - Research Facility, Whittier, California
  - Research Facility, Yuba City, California
  - Research Facility, Westminster, Colorado
  - Research Facility, Lauderdale Lakes, Florida
  - Research Facility, Miami, Florida
  - Research Facility, Pinecrest, Florida
  - Research Facility, Flossmoor, Illinois
  - Research Facility, Hines, Illinois
  - Research Facility, Louisville, Kentucky
  - Research Facility, Rockville, Maryland
  - Research Facility, Springfield, Massachusetts
  - Research Facility, Detroit, Michigan
  - Research Facility, Brookhaven, Mississippi
  - Research Facility, Brooklyn, New York
  - Research Facility, Flushing, New York
  - Research Facility, The Bronx, New York
  - Research Facility, Asheville, North Carolina
  - Research Facility, Toledo, Ohio
  - Research Facility, Oklahoma City, Oklahoma
  - Research Facility, Erie, Pennsylvania
  - Research Facility, Philadelphia, Pennsylvania
  - Research Facility, Providence, Rhode Island
  - Research Facility, Orangeburg, South Carolina
  - Research Facility, Arlington, Texas
  - Research Facility, Houston, Texas
  - Research Facility, San Antonio, Texas
  - Research Facility, Fairfax, Virginia
- Bulgaria (9):
  - Research Facility, Burgas
  - Research Facility, Pazardzhik
  - Research Facility, Pleven
  - Research Facility, Plovdiv
  - Research Facility, Rousse
  - Research Facility, Sofia
  - Research Facilities (2), Sofia
  - Research Facility, Varna
  - Research Facility, Veliko Tarnovo
- France (4):
  - Research Facility, Amiens
  - Research Facility, Bordeaux
  - Research Facility, Montpellier
  - Research Facility, Vannes
- Germany (4):
  - Research Facilities (2), Bremen
  - Research Facility, Franfurt
  - Research Facility, Hamburg
  - Research Facility, Kaiserslautern
- Italy (5):
  - Research Facility, Como
  - Research Facility, Cremona
  - Research Facility, Lecco
  - Research Facility, Modena
  - Research Facility, Prato
- Poland (4):
  - Research Facility, Ciechanów
  - Research Facility, Katowice
  - Research Facility, Pabianice
  - Research Facility, Włocławek
- Romania (2):
  - Research Facility, Bucharest
  - Research Facility, Iași
- Spain (5):
  - Research Facility, Alicante
  - Research Facility, Barcelona
  - Research Facility, Ciudad Real
  - Research Facility, Madrid
  - Research Facility, Santander
- United Kingdom (3):
  - Research Facility, Carshalton
  - Research Facility, London
  - Research Facility, Swansea

REFERENCES:
- [Result] Fishbane S, Schiller B, Locatelli F, Covic AC, Provenzano R, Wiecek A, Levin NW, Kaplan M, Macdougall IC, Francisco C, Mayo MR, Polu KR, Duliege AM, Besarab A; EMERALD Study Groups. Peginesatide in patients with anemia undergoing hemodialysis. N Engl J Med. 2013 Jan 24;368(4):307-19. doi: 10.1056/NEJMoa1203165. PMID 23343061
- [Derived] Macdougall IC, Provenzano R, Sharma A, Spinowitz BS, Schmidt RJ, Pergola PE, Zabaneh RI, Tong-Starksen S, Mayo MR, Tang H, Polu KR, Duliege AM, Fishbane S; PEARL Study Groups. Peginesatide for anemia in patients with chronic kidney disease not receiving dialysis. N Engl J Med. 2013 Jan 24;368(4):320-32. doi: 10.1056/NEJMoa1203166. PMID 23343062

RESULTS

PARTICIPANT FLOW:
Groups:
- Peginesatide: Participants received peginesatide by intravenous (IV) or subcutaneous (SC) injection once every 4 weeks. The starting dose was based on the participant's total weekly epoetin alfa or beta dose during the last week of the Screening Period; the first dose was administered one week after the last epoetin alfa or beta dose. Participants who received epoetin alfa or beta IV at the time of screening received peginesatide IV during the study, and participants who received epoetin alfa or beta SC at the time of screening received peginesatide SC during the study.
  The dose was adjusted to maintain hemoglobin levels in a target range of 10.0-12.0 grams per deciliter (g/dL) and ± 1.5 g/dL from baseline during the Titration and Evaluation Periods, and 10.0-12.0 g/dL during the Long-Term Safety and Efficacy Period.
- Epoetin: Participants continued to receive commercially available epoetin alfa or beta by intravenous or subcutaneous injection, at the same starting dose, frequency and route of administration as received during the last week of the Screening Period, with the first study dose of epoetin alfa or beta administered after randomization at Week 0.
  The dose was adjusted to maintain hemoglobin levels in a target range of 10.0-12.0 g/dL and ± 1.5 g/dL from baseline during the Titration and Evaluation Periods, and 10.0-12.0 g/dL during the Long-Term Safety and Efficacy Period.
Period: Overall Study
Arm/Group | Peginesatide | Epoetin
Started | 549 (Randomization was 2:1 peginesatide to epoetin) | 274
Completed | 421 | 211
Not Completed | 128 | 63
Not completed — Adverse Event | 4 | 2
Not completed — Death | 53 | 30
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 2 | 4
Not completed — Physician Decision | 3 | 0
Not completed — Pregnancy | 2 | 0
Not completed — Withdrawal by Subject | 44 | 12
Not completed — Discontinued Dialysis | 0 | 1
Not completed — Lost ability to consent | 1 | 1
Not completed — Never dosed | 1 | 0
Not completed — Relocation | 8 | 6
Not completed — Renal transplant | 9 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peginesatide | Epoetin | Total
Number analyzed (Participants) | 542 | 273 | 815
Age, Categorical [Count of Participants; unit: Participants] — Eight participants were excluded from the full analysis population: 7 participants in the Peginesatide group and 1 participant in the Epoetin group. These 8 participants did not receive study medication.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 350 | 173 | 523
    >=65 years | 192 | 100 | 292
Age Continuous [Mean (Standard Deviation); unit: years] | 58.8 (14.47) | 58.6 (13.73) | 58.8 (14.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 211 | 120 | 331
  Male | 331 | 153 | 484

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Hemoglobin Between Baseline and the Evaluation Period
Description: The baseline hemoglobin value is defined as the mean of five hemoglobin values: the four most recent hemoglobin values taken prior to the day of randomization and the value obtained on the day of randomization. The mean hemoglobin during the Evaluation Period for each participant is calculated as the mean of the available hemoglobin values during study Weeks 29 through 36.
Time Frame: Baseline to Weeks 29-36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Peginesatide | Epoetin
Number analyzed (Participants) | 542 | 273
g/dL
  Baseline [N=542, 273] | 11.20 (0.553) | 11.21 (0.546)
  Evaluation Period [N=488, 237] | 11.13 (1.018) | 11.05 (0.958)
  Change from Baseline [N=488, 237] | -0.07 (1.009) | -0.17 (1.000)
Statistical Analysis 1: Comparison: Peginesatide vs Epoetin; The sample size for this study has been determined based on a two group evaluation of non-inferiority using the t-distribution (one-sided significance level 0.025) with a non inferiority margin of -1.0 g/dL. A sample size of approximately 750 (peginesatide group of 500 and epoetin group of 250) provided at least 99% power for the evaluation of non-inferiority, assuming an expected treatment difference of 0.0 g/dL and a standard deviation of 1.5 g/dL; Test type: Non-Inferiority or Equivalence — A non-inferiority margin of -1.0 g/dL was used in the primary efficacy assessments. Non-inferiority was established if the lower limit of the two-sided 95% confidence interval for the difference between the means of the primary endpoint (peginesatide minus control ESA) was ≥ -1.0 g/dL; ANOVA; The ANOVA cell means model was used to estimate primary efficacy endpoint within the specified cells formed by the combination of treatment and strata; Least Squares Mean Difference = 0.10, 95% CI 2-sided [-0.05 to 0.26], Standard Error of Mean 0.078

2. Secondary Outcome: Proportion of Participants Who Receive Red Blood Cell (RBC) Transfusions During the Titration and Evaluation Periods
Time Frame: Weeks 0 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide | Epoetin
Number analyzed (Participants) | 542 | 273
percentage of participants | 0.077 | 0.099
Statistical Analysis 1: Comparison: Peginesatide vs Epoetin; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.79, 95% CI 2-sided [0.50 to 1.24]

3. Secondary Outcome: Proportion of Participants Whose Mean Hemoglobin Level During the Evaluation Period is Within the Target Range of 10.0 - 12.0 Grams Per Deciliter (g/dL)
Time Frame: Weeks 29 to 36
Population: Full Analysis Population: All randomized participants who received at least one dose of study medication
Measure: Number; unit: percentage of participants
Arm/Group | Peginesatide | Epoetin
Number analyzed (Participants) | 542 | 273
percentage of participants | 0.635 | 0.659
Statistical Analysis 1: Comparison: Peginesatide vs Epoetin; Test type: Superiority or Other; Cochran-Mantel-Haenszel; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.87 to 1.07]

ADVERSE EVENTS:
Arm/Group | Peginesatide | Epoetin
Serious Adverse Events (participants affected / at risk) | 268/542 | 141/273
Other Adverse Events (participants affected / at risk) | 445/542 | 222/273
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=542) | Epoetin (N=273)
Anaemia (Blood and lymphatic system disorders) | 5 | 5
Coagulopathy (Blood and lymphatic system disorders) | 2 | 1
Hypoprothrombinaemia (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 24 | 17
Acute myocardial infarction (Cardiac disorders) | 11 | 9
Cardiac arrest (Cardiac disorders) | 8 | 9
Atrial fibrillation (Cardiac disorders) | 8 | 8
Coronary artery disease (Cardiac disorders) | 8 | 7
Myocardial infarction (Cardiac disorders) | 10 | 4
Angina pectoris (Cardiac disorders) | 7 | 2
Cardio-respiratory arrest (Cardiac disorders) | 4 | 3
Bradycardia (Cardiac disorders) | 5 | 1
Cardiac failure (Cardiac disorders) | 4 | 2
Angina unstable (Cardiac disorders) | 3 | 2
Arrhythmia (Cardiac disorders) | 3 | 1
Sick sinus syndrome (Cardiac disorders) | 1 | 3
Acute coronary syndrome (Cardiac disorders) | 2 | 1
Pericarditis (Cardiac disorders) | 1 | 2
Supraventricular tachycardia (Cardiac disorders) | 2 | 1
Atrial flutter (Cardiac disorders) | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 1
Atrioventricular block complete (Cardiac disorders) | 2 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Nodal arrhythmia (Cardiac disorders) | 2 | 0
Tachycardia (Cardiac disorders) | 0 | 2
Aortic valve stenosis (Cardiac disorders) | 0 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 1 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 1 | 0
Dilatation ventricular (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve disease (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis uraemic (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Congenital cystic kidney disease (Congenital, familial and genetic disorders) | 1 | 0
Hyperparathyroidism (Endocrine disorders) | 2 | 0
Hyperparathyroidism secondary (Endocrine disorders) | 0 | 1
Hyperparathyroidism tertiary (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Vision blurred (Eye disorders) | 0 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 9 | 4
Gastritis erosive (Gastrointestinal disorders) | 4 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 1
Ascites (Gastrointestinal disorders) | 1 | 2
Colitis (Gastrointestinal disorders) | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 2 | 1
Appendicitis perforated (Gastrointestinal disorders) | 1 | 1
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 0
Large intestinal ulcer (Gastrointestinal disorders) | 1 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Erosive oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis atrophic (Gastrointestinal disorders) | 1 | 0
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gingivitis ulcerative (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal angina (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0
Oesophagitis ulcerative (Gastrointestinal disorders) | 1 | 0
Peptic ulcer perforation (Gastrointestinal disorders) | 1 | 0
Peritonitis (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 10 | 4
Chest pain (General disorders) | 8 | 5
Pyrexia (General disorders) | 2 | 5
Death (General disorders) | 3 | 2
Asthenia (General disorders) | 3 | 1
Catheter related complication (General disorders) | 1 | 2
Catheter thrombosis (General disorders) | 2 | 1
Chills (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Generalised oedema (General disorders) | 0 | 1
Ischaemic ulcer (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 3 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Anaphylactic shock (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 31 | 12
Sepsis (Infections and infestations) | 20 | 13
Cellulitis (Infections and infestations) | 19 | 5
Gastroenteritis (Infections and infestations) | 6 | 4
Bacteraemia (Infections and infestations) | 7 | 2
Urinary tract infection (Infections and infestations) | 7 | 1
Bronchitis (Infections and infestations) | 5 | 2
Osteomyelitis (Infections and infestations) | 4 | 3
Catheter related infection (Infections and infestations) | 4 | 2
Gangrene (Infections and infestations) | 4 | 2
Arteriovenous fistula site infection (Infections and infestations) | 2 | 3
Clostridium difficile colitis (Infections and infestations) | 5 | 0
Septic shock (Infections and infestations) | 2 | 3
Bronchopneumonia (Infections and infestations) | 2 | 2
Localised infection (Infections and infestations) | 2 | 2
Arteriovenous graft site infection (Infections and infestations) | 2 | 1
Pneumonia staphylococcal (Infections and infestations) | 1 | 2
Staphylococcal bacteraemia (Infections and infestations) | 2 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 2
Wound infection staphylococcal (Infections and infestations) | 1 | 2
Abdominal abscess (Infections and infestations) | 1 | 1
Abscess (Infections and infestations) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 2
Arthritis infective (Infections and infestations) | 2 | 0
Clostridium difficile sepsis (Infections and infestations) | 2 | 0
Diabetic foot infection (Infections and infestations) | 2 | 0
Diverticulitis (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 1
Enterococcal sepsis (Infections and infestations) | 2 | 0
Hepatitis B (Infections and infestations) | 2 | 0
Influenza (Infections and infestations) | 2 | 0
Lobar pneumonia (Infections and infestations) | 1 | 1
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 1
Osteomyelitis chronic (Infections and infestations) | 1 | 1
Pyelonephritis chronic (Infections and infestations) | 0 | 2
Sepsis syndrome (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1
Abscess limb (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 0 | 1
Bronchitis bacterial (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 1 | 0
Diabetic gangrene (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Incision site infection (Infections and infestations) | 1 | 0
Infected skin ulcer (Infections and infestations) | 0 | 1
Klebsiella bacteraemia (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Mastoiditis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Perinephric abscess (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Post procedural sepsis (Infections and infestations) | 1 | 0
Postoperative abscess (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Tuberculous pleurisy (Infections and infestations) | 0 | 1
Viraemia (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 10 | 6
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 5 | 2
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1 | 5
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3 | 3
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 4 | 1
Hip fracture (Injury, poisoning and procedural complications) | 3 | 2
Vascular graft complication (Injury, poisoning and procedural complications) | 4 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 3
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 3 | 0
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 3 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 | 0
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 2
Therapeutic product contamination (Injury, poisoning and procedural complications) | 2 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Delayed recovery from anaesthesia (Injury, poisoning and procedural complications) | 1 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0
Operative haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Procedural vomiting (Injury, poisoning and procedural complications) | 1 | 0
Renal haematoma (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Transplant failure (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Urinary anastomotic leak (Injury, poisoning and procedural complications) | 1 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Blood pressure increased (Investigations) | 1 | 0
Cardiac enzymes increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 25 | 8
Fluid overload (Metabolism and nutrition disorders) | 20 | 9
Hypoglycaemia (Metabolism and nutrition disorders) | 8 | 6
Diabetic foot (Metabolism and nutrition disorders) | 4 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 3 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Diabetic amyotrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 11 | 4
Syncope (Nervous system disorders) | 5 | 2
Convulsion (Nervous system disorders) | 3 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 3
Anoxic encephalopathy (Nervous system disorders) | 2 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 2
Cerebral infarction (Nervous system disorders) | 2 | 0
Encephalopathy (Nervous system disorders) | 2 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 2 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 2
Brain oedema (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebral haematoma (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Diabetic autonomic neuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Embolic stroke (Nervous system disorders) | 0 | 1
Facial palsy (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Hypoxic encephalopathy (Nervous system disorders) | 1 | 0
IIIrd nerve paralysis (Nervous system disorders) | 1 | 0
Intracranial aneurysm (Nervous system disorders) | 1 | 0
Myelopathy (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Syncope vasovagal (Nervous system disorders) | 0 | 1
Tardive dyskinesia (Nervous system disorders) | 1 | 0
Thrombotic stroke (Nervous system disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Mental status changes (Psychiatric disorders) | 5 | 3
Acute psychosis (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Hallucination (Psychiatric disorders) | 1 | 0
Azotaemia (Renal and urinary disorders) | 2 | 1
Renal failure chronic (Renal and urinary disorders) | 3 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0
Pyuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal haemorrhage (Renal and urinary disorders) | 1 | 0
Ureteric dilatation (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Urinary tract inflammation (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Penile necrosis (Reproductive system and breast disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Dry gangrene (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 11 | 3
Hypertensive crisis (Vascular disorders) | 8 | 4
Hypertension (Vascular disorders) | 3 | 3
Deep vein thrombosis (Vascular disorders) | 4 | 1
Malignant hypertension (Vascular disorders) | 2 | 3
Arteriosclerosis (Vascular disorders) | 2 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 1
Peripheral ischaemia (Vascular disorders) | 2 | 1
Peripheral vascular disorder (Vascular disorders) | 3 | 0
Hypertensive emergency (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arterial thrombosis limb (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0
Embolism (Vascular disorders) | 1 | 0
Extremity necrosis (Vascular disorders) | 1 | 0
Femoral artery occlusion (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Lymphocele (Vascular disorders) | 1 | 0
Lymphoedema (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Steal syndrome (Vascular disorders) | 0 | 1
Superior vena caval occlusion (Vascular disorders) | 0 | 1
Vascular pseudoaneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Peginesatide (N=542) | Epoetin (N=273)
Nausea (Gastrointestinal disorders) | 96 | 54
Diarrhoea (Gastrointestinal disorders) | 91 | 47
Vomiting (Gastrointestinal disorders) | 74 | 38
Constipation (Gastrointestinal disorders) | 56 | 27
Abdominal pain (Gastrointestinal disorders) | 51 | 21
Abdominal pain upper (Gastrointestinal disorders) | 29 | 11
Pyrexia (General disorders) | 61 | 29
Oedema peripheral (General disorders) | 53 | 18
Chest pain (General disorders) | 43 | 16
Asthenia (General disorders) | 41 | 12
Fatigue (General disorders) | 39 | 21
Pain (General disorders) | 30 | 10
Upper respiratory tract infection (Infections and infestations) | 53 | 24
Nasopharyngitis (Infections and infestations) | 46 | 24
Urinary tract infection (Infections and infestations) | 21 | 15
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 90 | 40
Procedural hypotension (Injury, poisoning and procedural complications) | 82 | 43
Vascular graft complication (Injury, poisoning and procedural complications) | 46 | 19
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 42 | 21
Procedural hypertension (Injury, poisoning and procedural complications) | 36 | 17
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 33 | 16
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 30 | 19
Fall (Injury, poisoning and procedural complications) | 30 | 11
Hyperkalaemia (Metabolism and nutrition disorders) | 41 | 16
Muscle spasms (Musculoskeletal and connective tissue disorders) | 106 | 52
Arthralgia (Musculoskeletal and connective tissue disorders) | 63 | 27
Back pain (Musculoskeletal and connective tissue disorders) | 61 | 23
Pain in extremity (Musculoskeletal and connective tissue disorders) | 61 | 36
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 34 | 15
Headache (Nervous system disorders) | 86 | 46
Dizziness (Nervous system disorders) | 43 | 25
Insomnia (Psychiatric disorders) | 38 | 23
Anxiety (Psychiatric disorders) | 28 | 23
Depression (Psychiatric disorders) | 23 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 96 | 50
Cough (Respiratory, thoracic and mediastinal disorders) | 69 | 35
Pruritus (Skin and subcutaneous tissue disorders) | 36 | 16
Hypertension (Vascular disorders) | 84 | 31
Hypotension (Vascular disorders) | 72 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first publication of the primary safety and efficacy results will include data from all appropriate study sites. Either after the first multicenter publication, or following 36 months after the completion of the study, Investigators are free to publish; such publications may not contain Sponsor Confidential Information and may be subject to Sponsor review 60 days prior to submission for publication.